CLINICAL TRIAL: NCT06148415
Title: Evaluation of Prenatal Attachment Levels and Spousal Adjustment in Couples Performing Fetal Heartbeat Monitoring
Brief Title: The Effect of Fetal Heartbeat Monitoring on Prenatal Attachment and Partner Adjustment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KSUESRAKARATASOKYAY004
Record Dates: First submitted 2023-11-18; First posted 2023-11-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy Related
Keywords: Attachment; Fetal Heart Sound; Partner compatibility

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial conducted with experimental and control groups.
Who Masked: Participant
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fetal Heartbeat Monitoring Group (Experimental): The prospective fathers will be trained by the investigators on how to perform the 1st and 2nd leopold maneuvers using visual materials. Each couple will be provided with a stethoscope to listen to the fetal heartbeat and will be given a schedule to listen to the fetal heartbeat together for 5-10 minutes at least once a day for 15 days.
  1. Leopold maneuver (Posture): The first maneuver is performed to determine the height of the fundus and the part that is located on the fundus.
  2. Leopold's maneuver (Position: back right, back left): This maneuver is used to determine which side the fetal back is on. On palpation, the side with the baby's back is flat and firmer, and the other side feels bumpy.
  Interventions: Behavioral: Fetal Heartbeat Monitoring Group
- Control (No Intervention): Standard care group without fetal heart rate monitoring

INTERVENTIONS:
Behavioral: Fetal Heartbeat Monitoring Group — Fetal Heartbeat Monitoring Group
  Arms: Fetal Heartbeat Monitoring Group

SUMMARY:
The aim of this interventional study is to obtain information about determining the effect of the following drugs. To evaluate prenatal attachment levels and spousal adjustment in couples with fetal heart rate monitoring.

The main questions it aims to answer are:

* Does fetal heart rate monitoring affect the attachment of pregnant women?
* Does fetal heart rate monitoring affect fathers' attachment?
* Does fetal heart rate monitoring affect pregnant women's adjustment to motherhood?

DETAILED DESCRIPTION:
Data will be collected from women who meet the inclusion criteria and agree to participate in the study. Data collection tools will be collected in 2 stages by the researcher using a questionnaire form by face-to-face interview method in a suitable room in previously determined hospitals.

In the first stage (Day 1); couples who meet the inclusion criteria will be informed about the study and written consent will be obtained from those who agree to participate in the study. The pre-test data collection phase will be completed by applying data collection tools. Then, the prospective fathers will be trained by the researchers on how to apply the 1st and 2nd leopold maneuvers using visual materials. Each couple will be provided with a stethoscope to listen to the fetal heartbeat, and they will be given a schedule to listen to the fetal heartbeat together for 5-10 minutes at least once a day for 15 days. During the training, the couples will be able to detect the fetal heartbeat in a healthy way and an appointment will be made for the second phase and the first phase of the study will be completed (approximately 10-15 minutes).

In the second phase (Day 15); the researchers will contact the women again and invite them to the ASM. Then, stethoscopes and charts will be received from the couples, data collection tools will be applied again and post-test data will be collected (1-5 minutes) and the data collection phase will be completed.

Pre-test data will be collected by applying data collection tools (Personal Information Form, Prenatal Self-Assessment Scale, Prenatal Mother Attachment Scale and Prenatal Father Attachment Scale) to the couples in the intervention group (Couples Monitoring Fetal Heartbeat) in the first interview. Then, the researchers will provide training on listening to the fetal heartbeat in the first stage and in the last session (Day 15), the data collection tools will be applied to the couples again and the post-test data will be collected and thus the data collection process will be completed.

No intervention will be applied to the women in the control group, however, in the first interview (Day 1), data collection forms (Personal Information Form, Prenatal Self-Assessment Scale, Prenatal Maternal Attachment Scale and Prenatal Paternal Attachment Scale) will be applied and pre-test data will be collected. Then, the post-test data will be collected by applying the data collection forms to the women again in the last session (Day 15) simultaneously with the application schedule in the experimental group and the data collection process will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate,
* Primigravida,
* Over 18 years of age,
* 32 weeks of gestation and above and without any diagnosed risk (such as pre-eclampsia, diabetes, heart disease, placenta previa, oligohydramnios, multiple pregnancy) in the current pregnancy,
* Those who do not have any diagnosed problems related to the health of the fetus (such as fetal anomaly, intrauterine growth retardation) will be included in the study.

Exclusion Criteria:

* Separated from his wife,
* In the first trimester of pregnancy,
* Those with any diagnosed risk in the mother or baby will not be included in the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of prenatal maternal attachment level | The Prenatal Maternal Attachment Scale will be administered to all pregnant women in both groups at the first interview (day 1).
  The scale has 19 items in total and each item focuses on the feelings, attitudes and behaviors of the pregnant woman towards the fetus. The scale is Likert-type and each item is scored between 1-5 (5= represents very strong feelings towards the fetus; 1= represents the absence of feelings towards the fetus). There are two sub-dimensions in the scale. The quality of attachment subscale refers to the quality of the pregnant woman's emotional experience of the fetus. The second sub-dimension, time spent on attachment, refers to the intensity of the time the pregnant woman spends thinking, talking and touching the fetus. A high score obtained from the scale indicates a high degree of attachment.
Assessment of prenatal maternal attachment level | Prenatal Maternal Attachment Scale will be administered to all pregnant women in both groups at the last interview (day 15).
  The scale has 19 items in total and each item focuses on the feelings, attitudes and behaviors of the pregnant woman towards the fetus. The scale is Likert-type and each item is scored between 1-5 (5= represents very strong feelings towards the fetus; 1= represents the absence of feelings towards the fetus). There are two sub-dimensions in the scale. The quality of attachment subscale refers to the quality of the pregnant woman's emotional experience of the fetus. The second sub-dimension, time spent on attachment, refers to the intensity of the time the pregnant woman spends thinking, talking and touching the fetus. A high score obtained from the scale indicates a high degree of attachment.
Assessment of prenatal paternal attachment level | The Prenatal Father Attachment Scale will be administered to all expectant fathers in both groups at the first interview (day 1).
  The Prenatal Father Attachment Scale is based on measuring the father's feelings and thoughts towards the developing baby in the womb in line with the father's experiences in the last two weeks. There are 9 reverse items in the scale consisting of 16 items. Reverse items are scored by reversing them. The scale has 2 sub-dimensions: "quality of attachment (8 items)" and "time spent on attachment (8 items)". The items are scored between 1-5 and a minimum score of 16 and a maximum score of 80 is obtained from the scale. The higher the score obtained from the scale, the higher the prenatal attachment is considered to be.
Assessment of prenatal paternal attachment level | The Prenatal Father Attachment Scale will be administered to all prospective fathers in both groups in the last interview (day 15).
  The Prenatal Father Attachment Scale is based on measuring the father's feelings and thoughts towards the developing baby in the womb in line with the father's experiences in the last two weeks. There are 9 reverse items in the scale consisting of 16 items. Reverse items are scored by reversing them. The scale has 2 sub-dimensions: "quality of attachment (8 items)" and "time spent on attachment (8 items)". The items are scored between 1-5 and a minimum score of 16 and a maximum score of 80 is obtained from the scale. The higher the score obtained from the scale, the higher the prenatal attachment is considered to be.
Assessment of spousal adjustment of pregnant women | Prenatal Self-Assessment Scale will be administered to all pregnant women in both groups in the first interview (day 1).
  This four-point Likert-type scale consists of 79 items. The scale has seven sub-dimensions: thoughts about her own and her baby's health, acceptance of pregnancy, acceptance of the maternal role, readiness for childbirth, fear of childbirth, relationship status with her own mother and relationship status with her partner. Each subscale contains between 10-15 items. Each item in the scale is evaluated on a four-point scale, and adaptation to pregnancy is scored from 1 to 4 (4: Very much defines, 3: Partially defines, 2: Somewhat defines, 1: Does not define at all). In this study, the relationship with spouse sub-dimension of the scale was used.
Assessment of spousal adjustment of pregnant women | Prenatal Self-Assessment Scale will be administered to all pregnant women in both groups at the last interview (day 15).
  This four-point Likert-type scale consists of 79 items. The scale has seven sub-dimensions: thoughts about her own and her baby's health, acceptance of pregnancy, acceptance of the maternal role, readiness for childbirth, fear of childbirth, relationship status with her own mother and relationship status with her partner. Each subscale contains between 10-15 items. Each item in the scale is evaluated on a four-point scale, and adaptation to pregnancy is scored from 1 to 4 (4: Very much defines, 3: Partially defines, 2: Somewhat defines, 1: Does not define at all). In this study, the relationship with spouse sub-dimension of the scale was used.

CONTACTS AND LOCATIONS:
Overall Officials: Esra KARATAŞ OKYAY, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared.

REFERENCES:
- [Background] Guney E, Ucar T. Effect of the fetal movement count on maternal-fetal attachment. Jpn J Nurs Sci. 2019 Jan;16(1):71-79. doi: 10.1111/jjns.12214. Epub 2018 May 17. PMID 29774647
- See also: Description citation link — https://pubmed.ncbi.nlm.nih.gov/29774647/